CLINICAL TRIAL: NCT04852848
Title: Creating a Sustainable Infrastructure for SARS-COV-2 (COVID-19) Testing at Syringe Exchange Programs
Brief Title: Creating a Sustainable Infrastructure for SARS-CoV-2 Testing (COVID-19) at Syringe Exchange Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11162020.013; 3R01DA037628-05S1 (NIH)
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-06

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect2Test Intervention (Experimental): A brief MI intervention to motivate individuals to participate in COVID-19 testing after receiving syringe exchange services
  Interventions: Behavioral: Connect2Test Intervention
- Control (No Intervention): Services as usual

INTERVENTIONS:
Behavioral: Connect2Test Intervention — Brief assessment based feedback and motivational interviewing intervention
  Arms: Connect2Test Intervention

SUMMARY:
PWIDs have been an underserved population in the context of the current pandemic; thus, little is known about the prevalence of COVID-19 and the acceptability and possible reach of testing for COVID-19 among PWIDs. To address this gap, this study leverages a current partnership with HIV Alliance (HIVA) in Oregon and our Community and Scientific Advisory Board to support implementation and sustainability of a COVID-19 testing program. Specifically, we will use community-based participatory approaches to develop, implement, and evaluate a COVID-19 testing program offered through HIVA's Syringe Services Programs (SSP), a natural point of care for PWIDs. The COVID-19 testing program will include procedures for sample collection, transmission of specimens to the University of Oregon CLIA-certified laboratory, and results reporting. Our clinical trial is a randomized control trial focused improving the uptake of testing through a motivational enhancement intervention: Connect2Test.

DETAILED DESCRIPTION:
People who inject drugs (PWIDs) are a socially vulnerable population and are exposed to risk factors including unstable housing and underlying medical conditions such as human immunodeficiency virus (HIV), tuberculosis (TB), and viral hepatitis that put them at increased risk for severe COVID-19 symptoms, including death. PWIDs also experience barriers such as a history of stigmatization and discrimination by health care systems and exposure to misinformation about testing that reduces access to health care services and testing. Because timely receipt of services relative to symptoms onset is critical for positive health outcomes and to reduce SARS-CoV-2 transmission, lack of testing has significant implications for PWID, highlighting an urgent need to increase testing uptake among this population. Despite this, PWIDs have been an underserved population in the context of the current pandemic; thus, little is known about the prevalence of COVID-19 and the acceptability and possible reach of testing for COVID-19 among PWIDs. To address this gap, this study leverages a current partnership with HIV Alliance (HIVA) in Oregon and our Community and Scientific Advisory Board to support implementation and sustainability of a COVID-19 testing program. Specifically, we will use community-based participatory approaches to develop, implement, and evaluate a COVID-19 testing program offered through HIVA's Syringe Services Programs (SSP), a natural point of care for PWIDs. Moreover, SSPs may offer a natural venue for dissemination and delivery of a vaccine, once available. The COVID-19 testing program will include procedures for sample collection, transmission of specimens to the University of Oregon CLIA-certified laboratory, and results reporting. For aim 1, we will assess the testing program utilization. For aim 2, we will develop and test a brief motivational enhancement intervention to optimize testing utilization among PWIDs. Using a randomized control trial, we will evaluate intervention effects on utilization of COVID-19 testing resources. For aim 3, we will collect data from syringe exchange staff and key volunteers on program acceptability, feasibility, appropriateness, adoption, and implementation barriers and facilitators related to the testing program and intervention. The current project has the potential to enhance COVID-19 testing access and reach among a significantly underserved population who experience multiple risks that make it difficult to prevent SARS-CoV-2 exposure and transmission and who are at increased risk for severe COVID-19 symptoms, if they were to contract the disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and over
* Attend Syringe Services Program
* English speaking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share IPD in line with requirements and protocols put forth by the RADx-UP data coordinating center (CDCC)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share IPD in the timeline put forth by the RADx-UP data coordinating center (CDCC)
Access Criteria: We will share IPD in line with requirements and protocols put forth by the RADx-UP data coordinating center (CDCC)

REFERENCES:
- [Derived] Mauricio AM, Cioffi CC, Sanders AM, Kosty D, Fernandes L, Mueller MV, Stormshak EA. A mixed methods evaluation of a motivational enhancement intervention to increase SARS-CoV-2 testing among people experiencing houselessness and people who inject drugs. Psychol Serv. 2025 Nov;22(4):688-698. doi: 10.1037/ser0000939. Epub 2025 Mar 31. PMID 40167545

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Connect2Test Intervention | Control
Started | 105 | 100
Completed | 105 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Connect2Test Intervention | Control | Total
Number analyzed (Participants) | 105 | 100 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.6) | 42.9 (13.7) | 43.1 (18.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 65 | 60 | 125
  Woman | 29 | 28 | 57
  Other or Unknown | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 77 | 71 | 148
  Unknown or Not Reported | 17 | 17 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 7 | 12
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 1 | 5
  White | 64 | 59 | 123
  More than one race | 15 | 13 | 28
  Unknown or Not Reported | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 105 | 100 | 205
Participants Tested Previously for SARS-CoV-2 [Count of Participants; unit: Participants] — Participants were asked to report whether they had ever been tested before for SARS-CoV-2. Response choices were yes or no. The baseline report indicates individuals who responded, "yes".
  Participants | 78 | 66 | 144

OUTCOME MEASURES:

1. Primary Outcome: Individual Participation in COVID-19 Testing
Description: Binary outcome, yes/no participated in COVID-19 tested, reported by CLIA laboratory
Time Frame: Immediately post-intervention assessment of whether clients participated in COVID-19 testing following either the brief intervention or services as usual
Measure: Count of Participants; unit: Participants
Arm/Group | Connect2Test Intervention | Control
Number analyzed (Participants) | 105 | 100
Participants | 25 | 21
Statistical Analysis 1: Comparison: Connect2Test Intervention vs Control; Test type: Equivalence — In our original power calculation, we expected to randomly assign 200 individuals to the Connect2Test (n = 100) and control conditions (n = 100). Power calculations were conducted using G*Power assuming a two-tailed test with alpha = .05, power = .80, and an estimated COVID-19 testing rate in the Connect2Test condition of 20%. With these assumptions, the minimum detectable effect size (odds ratio) is 2.46, which corresponds to a moderate Cohen's d (0.49); p = .6298, Chi-squared; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.61 to 2.27] — The control condition was the reference category (Connect2Test intervention = 1, Control = 0)

ADVERSE EVENTS:
Time Frame: 1 day (single point in time)
Arm/Group | Connect2Test Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/100
Other Adverse Events (participants affected / at risk) | 0/105 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT04852848/Prot_002.pdf
  • Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04852848/SAP_003.pdf
  • Informed Consent Form (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT04852848/ICF_004.pdf